CLINICAL TRIAL: NCT06450821
Title: PROSpECT-PRIOR-2-CHEMO: A Feasibility RCT of Novel Dental Intervention PRIOR[Proactive Intensive Oral Review & Treatment] in Patients Scheduled for Chemotherapy for Myeloma-ASCT & Hematological Cancers to Mitigate Chemotherapy Complications
Brief Title: PROSpECT-PRIOR-2-CHEMO: PRIOR Dental Intervention Before Chemo to Reduce Chemotherapy Complications
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Sue Pavitt, Professor, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 296640
Record Dates: First submitted 2024-02-29; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Oncology; Periodontitis; Myeloma; Oral Mucositis; Febrile Neutropenia
MeSH Terms: conditions — Neoplasms; Periodontitis; Neoplasms, Plasma Cell; Stomatitis; Febrile Neutropenia | interventions — Lead; Therapeutics

STUDY DESIGN:
Intervention Model Description: The moderate and high-risk patients will then be randomised. Those randomised to the PRIOR intervention arm will be assessed in a consultant-led Restorative Dentistry department & treatment offered to stabilise primary dental diseases (periodontal disease, caries, and odontogenic infection). The treatment plan (by a dentist) will be delivered within the therapeutic window (the PRIOR window), defined as the period between MDT decision to offer ASCT/allo-SCT up to 7 days prior to commencement of CT for ASCT/allo-SCT. Participant treatment plans are highly personalised and therefore number of visits within the therapeutic window to deliver PRIOR are not strictly defined. PRIOR will aim to stabilise the oral health of the participant and remove obvious sources of oral health infection. Participant follow-up will monitor febrile event rate and OM incidence between groups, within the participant therapeutic window, defined as day one of SCT/CT+100 days.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Control Arm: NHS standard care pathway delivered.
- Intervention Arm (Experimental): Intervention Arm: Professional Oral Health Care (POHC) referred to as PRIOR [Proactive Intensive Oral Review & Treatment] prior to chemotherapy.
  Interventions: Procedure: PRIOR [Proactive Intensive Oral Review & Treatment]

INTERVENTIONS:
Procedure: PRIOR [Proactive Intensive Oral Review & Treatment] — Intervention Arm: Professional Oral Health Care (POHC) referred to as PRIOR [Proactive Intensive Oral Review & Treatment] prior to chemotherapy.
  Arms: Intervention Arm

SUMMARY:
The aim of this feasibility trial is to determine if it is safe and feasible to treat oral health diseases in people with haematological cancers before they start their chemotherapy to reduce complications and disruption to planned chemotherapy dose or schedule.

DETAILED DESCRIPTION:
PROSpECT PRIOR-2-CHEMO is a feasibility trial which will determine if it is safe and feasible to introduce a new oral health (OH) "PRIOR"(Pro-Active Intensive Oral Review and Treatment prior to chemotherapy) intervention for people with cancer, prior to receiving chemotherapy (CT). PRIOR is a novel interdisciplinary intervention that will be introduced into the current oncology pathway and mirrors the specialist Restorative Dental pathway for patients undergoing treatment for Head and Neck cancers. PRIOR is aimed to be delivered within the relatively short therapeutic window that oncology patients have before commencing their scheduled CT for 1) myeloma-ASCT, or 2) Haematological Allograft SCT . This feasibility phase is valuable to inform a definitive trial. The definitive trial would provide important efficacy and mechanistic understanding of the mitigation of CT adverse events (Aes), specifically life-threatening febrile episodes and painful oral mucositis (OM).

The oral microbiome homeostasis is affected by CT; infection risk is exacerbated by OM, and other dental conditions like periodontal disease (PD) that damage the mucosa, caries, and acute / chronic odontogenic abscesses that collectively predispose to systemic translocation of oral-derived bacteria. With about 35% of the adult population affected by moderate and 10-15% severe periodontitis the importance of improving oral health and reducing bacteria load and portals of entry before CT is logical but seldom undertaken.

Bacteria are responsible for the two most prevalent human oral biofilm-mediated diseases: dental caries and periodontitis. Periodontitis is a chronic disease caused by inflammatory reactions to gram negative anaerobic bacteria, resulting in irreversible destruction to oral hard and soft tissues. Local inflammation and tissue damage allow oral bacteria to enter the bloodstream. These Immunocompromised patients (such as those receiving CT) are highly susceptible to these invading pathogens which can manifest as life-threatening systemic infections. The risk of developing systemic infections may be associated with the severity of periodontitis (i.e. the total surface area of the ulcerated pocket epithelium) and the composition periodontal pocket microbiota composition. OM is also an inflammatory condition affecting the oral mucosa. OM is a CT-induced complication that not only affects patient's quality of life but also acts as a portal for oral microorganisms and inflammatory products to translocate into the systemic circulation via the ulcerated mucosa. Pre-existing poor oral and periodontal health is a significant risk factors for CT-induced febrile events, creating therapeutic opportunity.

Oral infection, especially periodontitis, may affect the course and pathogenesis of a number of systemic diseases, including cancer, diabetes, and rheumatoid arthritis. The definitive trial will be a hypothesis-driven, mechanistic trial to understand the novel PRIOR intervention vs current NHS standard of care. Specifically, how PRIOR may mitigate Aes across a range of cancer types and CT regimens. The definitive aim is to understand how PRIOR impacts the oral microbial load, the portal entry sites, and the relationship between the oral microbiome, dysbiosis and systemic infection. The investigators will knowledge transfer from mechanistic evaluation of PD in rheumatoid arthritis showing the oral and gut microbiomes were perturbed but partly normalized after treatment. PD shares common mechanisms of action infection/inflammation across several systemic diseases.

Clinical guidelines recommend seeking dental care prior to CT, this may include recommendation to seek dental care with a general dental practitioner (GDP, Primary care), but uptake is low and established care pathways are rare. Consequently, there has been little direct clinical observation by oncology teams of the value of including dental review; In part due to low advocacy by the oncology team, fuelled by little direct clinical observation of the value of including dental review. Patients report significant barriers to achieving dental care prior to CT including access to a GDP, lack of perceived need and logistical challenges.

Patients do not prioritise seeking dental services as they are unaware of the potential importance to their oncology outcomes. The approach is to provide a specialist consultant-led hospital dental team review mirroring the specialist Restorative Dental pathway undertaken by patients having Head and Neck cancer treatment. Specialist dental teams within a secondary care setting may be better placed to deliver inter-disciplinary care than a GDP due to the time limited therapeutic window (therapeutic window defined as the period between diagnosis and deliver of CT). This work is the first to address the clinical need across several cancer patient groups.

ELIGIBILITY:
Inclusion Criteria (mod-high/risk trial participants):

* Adults (≥ 18years) with scheduled Chemotherapy. Specifically, patients who meet the following diagnosis and treatment window requirements:

  * Myeloma- Autologous Stem Cell Transplantation (ASCT) before high-dose myeloablative CT.
  * Haematological cancers suitable for Allografts Stem Cell Transplant (SCT) before CT
* Moderate / High Oral Health Risk Assessment - any one of the following:

  * Clinical evidence of caries (2+ teeth)
  * Clinical evidence on soft and hard tissue examination of infection, sinus, swelling or tenderness
  * BPE code 3-4 in any remaining sextant
  * BPE code 1-2 with >30% BOP
* The patient is fully informed, has received PIS (patient information sheet) and considered during a 'cooling-off' period, is competent to consent, and is able to comply with minimum attendance requirements

Exclusion Criteria:

* Have a history of head and neck radiotherapy
* Have been treated with Denusomab, Bevacizumab, Sunitinib or Aflibercept within 9 months of the MDT date.
* Insufficient teeth [defined as <2]
* Are incapable of providing informed written consent
* Are unable to comply with minimum attendance requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants able to attend treatment sessions required for completion of treatment plan, within the defined chemotherapy therapeutic window. | 100 days from the date of commencement of chemotherapy (about 4 months from randomisation)
  Ability to deliver individualised planned PRIOR intervention within the defined chemotherapy therapeutic window (no less than 7 days before the start of ASCT/allo-SCT) - Number of patients able to attend sessions required by treatment plan

SECONDARY OUTCOMES:
Ability to recruit, recruitment rate and acceptability of randomisation | Prior to commencement of CT and 100 days after CT
  Patients identified by oncology team, suitable for treatment within allotted time frame.
  Number of participants identified by oncology team and enrolled onto intervention vs standard of care arm.
Patient compliance with dental referral and treatment plan | Prior to commencement of CT and 100 days after CT
  Attrition rates. Ability to complete treatment within desired timeframe. Patients may not attend appointments due to various factors e.g. illness, timing etc.
  Consent withdrawal from treatment, patients understanding of treatment etc.
  Measured by number of patients identified to number of participants who complete treatment
Ability to collect samples (baseline and febrile events) for trial biobank future oral biology testing/mechanistic evaluation | Prior to commencement of CT and 100 days after CT
  Baseline samples collected by dental team, febrile events collected by oncology team.
Data collection via electronic health records | Prior to commencement of CT and 100 days after CT
  E.g Oral mucositis and febrile events. Electronic health records accessed by dental team (with patients consent)
Number of participants developing sepsis/bloodstream infection/febrile events | 100 days after CT
  Feasibility of collecting clinical assessments from electronic health records /PROMS [This will also support primary outcome selections and inform power calculations assumptions for a definitive trial]
Number of participants developing oral mucositis and returning the OMDQ questionnaire | 100 days after CT
  Feasibility of collecting clinical assessments from electronic health records /PROMS [This will also support primary outcome selections and inform power calculations assumptions for a definitive trial]
Number of participants prescribed an Antibiotic | 100 days after CT
  Feasibility of collecting clinical assessments from electronic health records /PROMS [This will also support primary outcome selections and inform power calculations assumptions for a definitive trial]
Number of participants with hospital admissions and the length of their hospital stays | 100 days after CT
  Feasibility of collecting clinical assessments from electronic health records /PROMS [This will also support primary outcome selections and inform power calculations assumptions for a definitive trial]
Number of participants with other (specified) chemotherapy-related complications | 100 days after CT
  Feasibility of collecting clinical assessments from electronic health records /PROMS [This will also support primary outcome selections and inform power calculations assumptions for a definitive trial]
Number of participants completing Quality of Life Questionnaires | 100 days after CT
  (EORTC QLQ-C30; QLQ-OH15) Feasibility of collecting clinical assessments from electronic health records /PROMS [This will also support primary outcome selections and inform power calculations assumptions for a definitive trial]
Rate of Mortality | 100 days after CT
  Feasibility of collecting clinical assessments from electronic health records /PROMS [This will also support primary outcome selections and inform power calculations assumptions for a definitive trial]
Process Evaluation | post 100 days
  Acceptability of delivery of PRIOR to participants and clinical delivery teams in haematology and dental departments - Focus group/Interviews
Inform the design of a definitive RCT. Specifically, whether haematological cancer groups can be combined for efficiency | After completion of study, approximately 18 months
  Ability to perform a power calculation to inform a future trial the ideal number of sites required, to make informed decisions about stop/go progression criteria to monitor the trial's progress effectively.

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Ali, BChD, Principal Investigator — LTHT
Locations (1):
- Dental Translational & Clinical Research Unit (DenTCRU), Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Background] Raber-Durlacher JE, Epstein JB, Raber J, van Dissel JT, van Winkelhoff AJ, Guiot HF, van der Velden U. Periodontal infection in cancer patients treated with high-dose chemotherapy. Support Care Cancer. 2002 Sep;10(6):466-73. doi: 10.1007/s00520-002-0346-3. Epub 2002 Mar 23. PMID 12353125
- [Background] Brennan MT, Elting LS, Spijkervet FK. Systematic reviews of oral complications from cancer therapies, Oral Care Study Group, MASCC/ISOO: methodology and quality of the literature. Support Care Cancer. 2010 Aug;18(8):979-84. doi: 10.1007/s00520-010-0856-3. Epub 2010 Mar 20. PMID 20306090
- [Background] Jia G, Zhi A, Lai PFH, Wang G, Xia Y, Xiong Z, Zhang H, Che N, Ai L. The oral microbiota - a mechanistic role for systemic diseases. Br Dent J. 2018 Mar 23;224(6):447-455. doi: 10.1038/sj.bdj.2018.217. PMID 29569607
- [Background] Zecha JAEM, Raber-Durlacher JE, Laheij AMGA, Westermann AM, Epstein JB, de Lange J, Smeele LE. The impact of the oral cavity in febrile neutropenia and infectious complications in patients treated with myelosuppressive chemotherapy. Support Care Cancer. 2019 Oct;27(10):3667-3679. doi: 10.1007/s00520-019-04925-8. Epub 2019 Jun 20. PMID 31222393
- [Background] Laine PO, Lindqvist JC, Pyrhonen SO, Strand-Pettinen IM, Teerenhovi LM, Meurman JH. Oral infection as a reason for febrile episodes in lymphoma patients receiving cytostatic drugs. Eur J Cancer B Oral Oncol. 1992 Oct;28B(2):103-7. doi: 10.1016/0964-1955(92)90036-z. PMID 1306727
- [Background] Borowski B, Benhamou E, Pico JL, Laplanche A, Margainaud JP, Hayat M. Prevention of oral mucositis in patients treated with high-dose chemotherapy and bone marrow transplantation: a randomised controlled trial comparing two protocols of dental care. Eur J Cancer B Oral Oncol. 1994;30B(2):93-7. doi: 10.1016/0964-1955(94)90059-0. PMID 8032307
- [Background] Tsuji K, Shibuya Y, Akashi M, Furudoi S, Yakushijin K, Kawamoto S, Okamura A, Matsuoka H, Komori T. Prospective study of dental intervention for hematopoietic malignancy. J Dent Res. 2015 Feb;94(2):289-96. doi: 10.1177/0022034514561768. Epub 2014 Dec 10. PMID 25503612
- [Background] Zhang X, Zhang D, Jia H, Feng Q, Wang D, Liang D, Wu X, Li J, Tang L, Li Y, Lan Z, Chen B, Li Y, Zhong H, Xie H, Jie Z, Chen W, Tang S, Xu X, Wang X, Cai X, Liu S, Xia Y, Li J, Qiao X, Al-Aama JY, Chen H, Wang L, Wu QJ, Zhang F, Zheng W, Li Y, Zhang M, Luo G, Xue W, Xiao L, Li J, Chen W, Xu X, Yin Y, Yang H, Wang J, Kristiansen K, Liu L, Li T, Huang Q, Li Y, Wang J. The oral and gut microbiomes are perturbed in rheumatoid arthritis and partly normalized after treatment. Nat Med. 2015 Aug;21(8):895-905. doi: 10.1038/nm.3914. Epub 2015 Jul 27. PMID 26214836
- [Background] Momen-Heravi F, Babic A, Tworoger SS, Zhang L, Wu K, Smith-Warner SA, Ogino S, Chan AT, Meyerhardt J, Giovannucci E, Fuchs C, Cho E, Michaud DS, Stampfer MJ, Yu YH, Kim D, Zhang X. Periodontal disease, tooth loss and colorectal cancer risk: Results from the Nurses' Health Study. Int J Cancer. 2017 Feb 1;140(3):646-652. doi: 10.1002/ijc.30486. Epub 2016 Nov 23. PMID 27778343
- [Background] D'Aiuto F, Gkranias N, Bhowruth D, Khan T, Orlandi M, Suvan J, Masi S, Tsakos G, Hurel S, Hingorani AD, Donos N, Deanfield JE; TASTE Group. Systemic effects of periodontitis treatment in patients with type 2 diabetes: a 12 month, single-centre, investigator-masked, randomised trial. Lancet Diabetes Endocrinol. 2018 Dec;6(12):954-965. doi: 10.1016/S2213-8587(18)30038-X. Epub 2018 Oct 24. PMID 30472992
- [Background] Konig MF, Abusleme L, Reinholdt J, Palmer RJ, Teles RP, Sampson K, Rosen A, Nigrovic PA, Sokolove J, Giles JT, Moutsopoulos NM, Andrade F. Aggregatibacter actinomycetemcomitans-induced hypercitrullination links periodontal infection to autoimmunity in rheumatoid arthritis. Sci Transl Med. 2016 Dec 14;8(369):369ra176. doi: 10.1126/scitranslmed.aaj1921. PMID 27974664
- [Background] Keefe DM, Schubert MM, Elting LS, Sonis ST, Epstein JB, Raber-Durlacher JE, Migliorati CA, McGuire DB, Hutchins RD, Peterson DE; Mucositis Study Section of the Multinational Association of Supportive Care in Cancer and the International Society for Oral Oncology. Updated clinical practice guidelines for the prevention and treatment of mucositis. Cancer. 2007 Mar 1;109(5):820-31. doi: 10.1002/cncr.22484. PMID 17236223